CLINICAL TRIAL: NCT06533956
Title: Programme D'Entrainement À La Marche Avec Blood Flow RestrIctioN Chez L'enfant Avec Paralysie Cérébrale - EMBRIN: Etude Pilote
Brief Title: Gait Training Program with Blood Flow Restriction in Children with Cerebral Palsy - EMBRIN: Pilot Study
Acronym: EMBRIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49RC23_0258
Record Dates: First submitted 2024-07-23; First posted 2024-08-01 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Blood Flow Restriction; Walking training; Pediatric rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- gait training associated with BFR (Experimental): The children will receive a 10-week intervention (1 week of habituation without BFR + 9 weeks with BFR) comprising 3 30-minute treadmill sessions per week. At each session, the first 5 minutes will enable a gradual increase in speed, and then the maximum tolerated walking speed will be sought. Maximum speed corresponds to the walking speed maintained by the child for an effort of between 5 and 7 on Borg's 10-point VAS. The rehabilitator will encourage the child to maintain this speed and provide feedback on performance. The BFR setting will maintain an occlusion, at the root level of both lower limbs, of 60% of the total occlusal pressure.
  Interventions: Other: 10-week gait training program combined with simultaneous blood flow restriction (BFR).

INTERVENTIONS:
Other: 10-week gait training program combined with simultaneous blood flow restriction (BFR). — The children will receive a 10-week intervention (1 week of habituation without BFR + 9 weeks with BFR) comprising 3 30-minute treadmill sessions per week. At each session, the first 5 minutes will enable a gradual increase in speed, and then the maximum tolerated walking speed will be sought. Maximum speed corresponds to the walking speed maintained by the child for an effort of between 5 and 7 on Borg's 10-point VAS. The rehabilitator will encourage the child to maintain this speed and provide feedback on performance. The BFR setting will maintain an occlusion, at the root level of both lower limbs, of 60% of the total occlusal pressure.

SUMMARY:
This is a single-center prospective experimental pilot study to assess the feasibility, tolerability and effect of a 10-week gait training program combined with simultaneous blood flow restriction (BFR) on the walking speed of children, aged 8 to 18, with bilateral spastic cerebral palsy.

The children will receive a 10-week intervention (1 week of habituation without BFR + 9 weeks with BFR) comprising 3 30-minute treadmill sessions per week. At each session, the first 5 minutes will enable a gradual increase in speed, and then the maximum tolerated walking speed will be sought. Maximum speed corresponds to the walking speed maintained by the child for an effort of between 5 and 7 on Borg's 10-point VAS. The rehabilitator will encourage the child to maintain this speed and provide feedback on performance. The BFR setting will maintain an occlusion, at the root level of both lower limbs, of 60% of the total occlusal pressure.

Children receiving the 10-week EMBRIN program are expected to improve their walking ability and muscular strength, two targets recognized as priorities for individuals with CP by the HAS. In this population, a major limitation of implementing rehabilitation programs is the large amount of practice required to bring about significant changes. This large amount of practice requires a major investment on the part of the individual, as well as significant rehabilitation resources. Muscle-strengthening programs are also particularly repetitive and therefore not very motivating for children. The EMBRIN program could reduce the training load and duration required to impact functional performance in children with CP. It could also help reduce the cost of rehabilitation interventions and reduce physical therapy time for individuals with CP in favor of their social participation.

DETAILED DESCRIPTION:
Context :

Cerebral palsy (CP) is the leading cause of motor disability in children, with a prevalence of 1.77 cases per 1000 births. It is defined as a set of permanent developmental disorders of movement and posture, resulting from a non-progressive brain lesion affecting a developing brain. 60% of individuals with CP have a bilateral form. In this group, 98% of diplegics and 24% of quadriplegics will be "walkers", but more often than not with poor walking efficiency. In fact, these children show not only a reduction in walking speed, but also markedly reduced endurance. What's more, these children have reduced levels of physical activity, resulting in less participation in physical activities throughout their lives. Associated with these changes in motor activity, CP leads to morphological and architectural changes in the muscles, including reduced muscle volume, shorter muscle fascicles and increased intramuscular fat. These "bad" adaptations contribute to a reduction in muscle strength and power, leading to a progressive decline in functional capacity in adolescence and adulthood, associated with a sedentary lifestyle. In individuals with CP, gait training and muscle strengthening programs, carried out separately, have shown, respectively, a relative efficacy in improving walking activity and lower limb muscle strength. Rare programs combining these two interventions have been shown to be of interest in mildly affected children. In the geriatric population (without CP), where strengthening with heavy loads may be contraindicated and difficult to implement, Blood Flow Restriction (BFR) training has attracted considerable interest due to its simplicity of use and effectiveness. Indeed, the application of an inflatable cuff to the proximal part of a limb restricting blood flow, combined with low-load muscle strengthening, has shown similar effects to high-load strengthening on muscle function. BFR was also combined with functional training, and this combination showed superiority over functional training alone in improving functional activity. BFR does not appear to cause side-effects in typical adolescents, and has never been studied in children with CP.

Objectives and evaluation criteria :

Primary objective: to study the effect of a 10-week gait training program combined with simultaneous blood flow restriction (BFR), using a commercially available device, on the walking speed of children aged 8 to 18 with bilateral spastic cerebral palsy. To this end, a comparison of patients' walking speed will be carried out between the period D-70 to D0 (standard rehabilitation) and the period D0 to D+70 (walking training program + BFR). Walking speed will be assessed by the 10-meter walk test. The evaluation criterion is the change in walking speed between D-70-J0 and D0-J+70.

Secondary objectives and evaluation criteria

To assess the effect of this gait training program combined with BFR on the following levels of the International Classification of Functioning and Disability:

Functions :

* Isometric strength of plantar flexors, knee extended and flexed, by electronic hand dynamometer (DEM)
* Isometric strength of knee flexors and extensors by DEM
* Isometric strength of hip abductors by DEM
* Pain intensity by numerical rating scale (NRS-11) (somato sensory function)

Activities :

* Walking endurance by 6-minute walk test
* Spontaneous and maximum walking speeds using the 10-meter walk test
* Global motor activity via Gross Motor Function Measure - 66 (GMFM-66)
* Spatial gait parameters: stride length, step length, base of support, step angle, and temporal gait parameters: speed and normalized speed, cadence, percentage of right and left support phase, right and left cycle time and double support time (Gaitrite)

Participation:

* Achievement of functional goals in terms of performance and satisfaction using the Canadian Occupational Performance Measure (COPM)
* Achievement of daily activities and mobility using the Pediatric Evaluation of Disability Inventory as a computer adaptive test (PEDI-CAT)
* Evaluate the feasibility of this gait training program associated with BFR. Feasibility will be assessed by analyzing the percentage of children completing 80% of the training program.
* To evaluate the tolerance of the EMBRIN program of this gait training program associated with BFR. Tolerance to the training program will be studied by assessing pain before, during and after gait training with the NRS-11 scale (23), as well as by notifying the occurrence of intercurrent medical events or complications. The evaluation criteria are :
* Change in NRS-11 pain score during gait training sessions;
* The occurrence of intercurrent medical events or complications.
* Evaluate participant satisfaction using the CSQ-8 satisfaction questionnaire.

Research scheme and progress This is a single-center prospective experimental pilot study designed to assess the feasibility, tolerability and effect of a 10-week gait training program combined with simultaneous blood flow restriction (BFR) on the walking speed of children, aged 8 to 18, with bilateral spastic cerebral palsy. The children will receive a 10-week intervention (1 week of habituation without BFR + 9 weeks with BFR) comprising 3 30-minute treadmill sessions per week. At each session, the first 5 minutes will enable a gradual increase in speed, and then the maximum tolerated walking speed will be sought. Maximum speed corresponds to the walking speed maintained by the child for an effort of between 5 and 7 on Borg's 10-point VAS. The rehabilitator will encourage the child to maintain this speed and provide feedback on performance. The BFR setting will maintain an occlusion, at the root level of both lower limbs, of 60% of the total occlusal pressure.

During each session, pain will be assessed using the NRS-11 before the restriction is placed, after 15 minutes of walking and within 5 minutes of the restriction being removed. In the event of participant request or premature termination of the session, a pain assessment will be added. A pain assessment will also be carried out 24 hours after the training session.

Functional assessments carried out at baseline at T0 (D0-70d) and T1 (D0) will explore the usual evolution of walking speed in children receiving usual care. Assessments at T2 (D0+35d) will explore the evolution of variables of interest halfway through the intervention period. Evaluations at T3 (D0+70d) will assess the immediate effects of therapy. Functional assessments will be carried out again at T4 (D0+100d) and T5 (D0+160) to evaluate the medium-term effect of therapy.

Research duration Inclusion period: 24 months Duration of participation: 8 months maximum Study duration: 32 months

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 8 to 18 with bilateral spastic cerebral palsy
* Patient with functional level II or III according to the Gross Motor Function Classification System (GMFCS)
* Patient able to assess pain with NRS-11
* Patient able to walk on a treadmill without body weight support, with or without technical aids
* Patient able to perform the 10-meter walk test
* No skin pathology at the pressure cuff application site (eczema, inflammatory scarring, etc.)
* Patient affiliated to or benefiting from a social security scheme
* Informed consent, dated and signed by parents or guardians (if a minor) or by the patient (if of age), to participate in the study;

Exclusion Criteria:

* Patients who have undergone surgical treatment or intramuscular injections of botulinum toxin in the lower limbs within the last 3 months
* Patients with a history of arterial hypertension, thrombo-embolic events, thrombophilia or cancer.
* Patient with insufficient understanding of the French language;
* Opposition of the patient (child or adolescent);
* Pregnant, breast-feeding or parturient women;
* Persons deprived of their liberty by judicial or administrative decision;
* Persons under compulsory psychiatric care;
* Persons under legal protection

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of changes in walking speed with standard rehabilitation and with gait training associated with BFR. | Patients' walking speed will be compared between Day -70 to Day 0 (standard rehabilitation) and Day 0 to Day +70 (gait training program + BFR)
  The evaluation criterion is the change in walking speed between D-70-J0 and D0-J+70.

CONTACTS AND LOCATIONS:
Overall Officials: Adélie Christiaens, Principal Investigator — University Hospital, Angers
Locations (2):
- France (2):
  - Les Capucins, Angers
  - University Hospital, Angers, Angers

IPD SHARING:
Plan to Share IPD: No